CLINICAL TRIAL: NCT03514810
Title: Combined Sertraline and Ketoprofen Administration in Major Depressive Disorder
Acronym: Srt+ktpMDD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kufa University (Other)
Responsible Party: Principal Investigator, Hussein Kadhem Al-Hakeim, Professor, Kufa University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KufaU; Arafataldujaili (Other: College of Science)
Record Dates: First submitted 2018-04-13; First posted 2018-05-02 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder; sertraline; ketoprofen
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Ketoprofen; Sertraline; Interleukins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sertralin & Ketoprofen in MDD (Placebo Comparator): To compare the median of Beck Depression Inventory-II (BDI-II) score of MDD patients after treatment with sertralin (50mg) daily+placebo and after treatment with combination of (sertralin & ketoprofen) for two months.
  Interventions: Combination Product: Combined Sertraline & Ketoprofen; Other: Interleukins in MDD after treatment
- Interleukins in MDD after treatment (Experimental): Some Interleukines level were estimated before and after treatment with sertralin 50 mg in combination with either placebo or ketoprofen 100mg daily.
  Interventions: Combination Product: Combined Sertraline & Ketoprofen; Other: Interleukins in MDD after treatment

INTERVENTIONS:
Combination Product: Combined Sertraline & Ketoprofen — The first group of patients has administered sertralin (50mg)+placebo. The second group has administered sertralin (50mg)+ketoprofen (100mg) (Sertraline & Ketoprofen) daily.
  Other Names: Zoloft & Ketoprofen
Other: Interleukins in MDD after treatment — Some interleukine levels were estimated in the first group of patients (administered sertralin,50mg+ketoprofen,100mg) and compared with their level in the second group (administered sertralin (50mg)+placebo).
  Other Names: Effect Ketoprofen & Sertraline on MDD

SUMMARY:
Among the major depressive disorder (MDD) patients in the follow-up group, 16 were administered with 50 mg of oral sertralin once daily with placebo, whereas 28 were treated with 100 mg of ketoprofen once daily as adjuvant treatment for MDD. Controls do not take any medicine.

DETAILED DESCRIPTION:
The research is a prospective, 2-month, double-blind study of parallel groups of patients with MDD with or without ketoprofen administration in addition to sertralin.

1. Patients: A total of 140 patients with MDD (78 male and 62 female; aged 18-65 years) participated in the study. Two samples were obtained at the beginning and 2 months after treatment from 34 patients that were followed up for two months after treatment. The samples were collected from "The Psychiatry Unit" at Al-Hakeem General Hospital in Najaf Governorate-Iraq from November 2016 to August 2017. Patient samples were also obtained from a private psychiatric clinic that was run by an assistant professor in psychiatric medicine. The patients were diagnosed by psychiatrists in accordance with a semi-structured psychiatric interview schedule for MDD diagnosis based on the 10th revision of the International Statistical Classification of Diseases and Related Health Problems. The full medical histories of the patients were evaluated such that any existing systemic disease that may affect the parameters to be diagnosed, particularly diabetes, liver disease, and renal disease, were excluded. Patients with histories of these diseases were excluded from the study. Serum C-reactive protein (CRP) was negative in all of the samples (CRP<6 mg/L). This test was conducted to exclude the presence of any overt infection or inflammation that may elevate acute-phase-reactant proteins, especially CRP. The protocol was approved by the IRB of the University of Kufa. The patients or their close first-degree relatives provided informed consent in accordance with the procedures outlined by the current IRB.

   Among the patients in the follow-up group, 16 were administered with 50 mg of oral sertralin once daily with placebo, whereas 28 were treated with 100 mg of ketoprofen once daily as adjuvant treatment for MDD.
2. Controls: As part of the control group, 40 apparently healthy subjects (22 males and 18 females) were selected. Their sex and age were matched with those of the patients. These subjects were apparently free from psychiatric and somatic diseases.

ELIGIBILITY:
Inclusion Criteria:

* The patients were diagnosed by psychiatrists in accordance ICD10 as having major depressive disorder.
* The patients had no existing systemic disease that may affect the parameters to be diagnosed.
* Patients with negative serum C-reactive protein (CRP<6 mg/L).

Exclusion Criteria:

* Patients with any systemic disease particularly diabetes, liver disease, and renal disease
* Patients with positive CRP
* Patients who taking any other drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2017-09-10 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Reduction in the Beck Depression Inventory-II Score | 12 months
  BDI-II is a 21-item self-report scale measuring current depressive symptoms. The standardized cutoffs used differ from the original:
  * 0-13: minimal depression
  * 14-19: mild depression
  * 20-28: moderate depression
  * 29-63: severe depression. Reduction in the Beck Depression Inventory-II Score by Combined Sertraline and Ketoprofen Administration in Major Depressive Disorder

SECONDARY OUTCOMES:
Decrease in Serum of IL-1β, IL-6, and IL-18 Levels | 12 months
  Decrease in Serum of IL-1β, IL-6, and IL-18 Levels by Combined Sertraline and Ketoprofen Administration in Major Depressive Disorder.
  All these cytokines were measured using ng/ml unit.
Body mass index (BMI) | 2 months
  Body mass index (BMI) is a measure for obesity and low weight measure. It is chosen because the MDD patients have a change in appetite and monitoring the weight is importany indication of normal appetite and cure. BMI Categories:
  Underweight = <18.5 Normal weight = 18.5-24.9 Overweight = 25-29.9 Obesity = BMI of 30 or greater

CONTACTS AND LOCATIONS:
Overall Officials: Arafat H Al-dujaili, PhD, Principal Investigator — Head of Department of Psychiatry

IPD SHARING:
Plan to Share IPD: No
Direct contact on my e-mail:headm2010@yahoo.com